CLINICAL TRIAL: NCT04753489
Title: Randomized Crossover 2-Period Single-dose BE Study of Rivaroxaban Film-coated Tablets 10mg (Pharmtechnology LLC, Republic of Belarus) and Xarelto® Film-coated Tablets 10mg (Bayer AG, Germany) in Healthy Male Volunteers in Fasting Conditions
Brief Title: Bioequivalence Study of Two Formulations of Rivaroxaban Tablets 10 mg in Healthy Male Volunteers in Fasting Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: ClinPharmInvest, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: RVRX_10-2020-CPD-FRMT
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Bioequivalence
Keywords: Rivaroxaban; Bioequivalence; Xarelto

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence TR (Other): 17 subjects assigned to the sequence TR will receive a single 10 mg dose of the test product Rivaroxaban (1 x 10 mg tablet), marked as T in the sequence, in Period 1 and a single 10 mg dose of the reference product Xarelto® (1 x 10 mg tablet), marked as R in the sequence, in period 2. These treatments will be administered orally with approximately 200 mL of water, in the morning, after overnight fasting. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Rivaroxaban film-coated tablet 10 mg; Drug: Xarelto® film-coated tablet 10 mg
- Sequence RT (Other): 17 subjects assigned to the sequence RT will receive a single 10 mg dose of the reference product Xarelto® (1 x 10 mg tablet), marked as R in the sequence, in Period 1 and a single 10 mg dose of the test product Rivaroxaban (1 x 10 mg tablet), marked as T in the sequence, in period 2. These treatments will be administered orally with approximately 200 mL of water, in the morning, after overnight fasting. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Rivaroxaban film-coated tablet 10 mg; Drug: Xarelto® film-coated tablet 10 mg

INTERVENTIONS:
Drug: Rivaroxaban film-coated tablet 10 mg — Rivaroxaban is manufactured by Pharmtechnology LLC, Republic of Belarus. Each tablet contains 10 mg of rivaroxaban.
  Other Names: The test product
Drug: Xarelto® film-coated tablet 10 mg — Xarelto® is manufactured by Bayer AG, Germany. Each tablet contains 10 mg of rivaroxaban.
  Other Names: The reference product

SUMMARY:
This is an open-labeled, laboratory-blinded, randomized, two period, single-center, crossover, comparative study, where each participant will be randomly assigned to the reference (Xarelto®, 10 mg film-coated tablets) or the test (Rivaroxaban, 10 mg film-coated tablets) formulation in each period of study (sequences Test-Reference (TR) or Reference-Test (RT)), in order to evaluate if both formulations are bioequivalent.

ELIGIBILITY:
Inclusion Criteria:

1. healthy caucasian men aged between 18 to 45 years;
2. verified diagnosis "healthy" according to the anamnesis data and the results of standard clinical, laboratory and instrumental examination methods, physical examination and anamnestic examination;
3. body mass index 18.5-30 kg/m²;
4. the results of an X-ray or fluorographic examination of the chest organs within the normal range (the results of an examination carried out within 12 months before the start of the study may be provided);
5. consent to use a double barrier method of contraception (condom + spermicide) or complete sexual abstinence, as well as consent not to take part in sperm donation from the moment of taking the drug in the first period, during the entire study and within 14 days after taking the drug in the second period research;
6. subjects are able to understand the requirements of the study, to sign a written informed consent, and also to accept all the restrictions imposed during the course of the study, and to agree to return for the required investigations.

Exclusion Criteria:

1. burdened allergic history, hypersensitivity to rivaroxaban or excipients that are part of any of the investigational drugs, or intolerance to these components;
2. clinically significant pathologies of the cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract, liver, kidneys and blood;
3. other diseases that, in the opinion of the researcher, may affect the absorption, distribution, metabolism or excretion of both drugs, or increase the risk of negative consequences for the volunteer;
4. a history of brain or spinal cord injury, recent surgery on the brain, spinal cord or eyes;
5. history of internal bleeding of any genesis;
6. a history of coagulation disorders (eg, von Willebrand disease, hemophilia);
7. hereditary intolerance to lactose or galactose (for example, congenital lactase deficiency or glucose-galactose malabsorption), since the composition of the tested and reference drugs includes lactose monohydrate;
8. the presence of mental disorders, including a history;
9. seizures, epilepsy and any other neurological disorders in history;
10. surgical interventions on the gastrointestinal tract, with the exception of appendectomy;
11. acute infectious diseases that ended less than 4 weeks before taking the drug in the first period;
12. dehydration due to diarrhea, vomiting or other reason within the last 24 hours before taking the drug in the first period of the study. Moreover, if vomiting or diarrhea was a manifestation of an infectious disease, then participation in the study is possible only 4 weeks after the last symptom.
13. Clinically significant abnormalities on the ECG, the level of systolic blood pressure (SBP) measured in the sitting position at the time of screening <100 mm Hg or ≥ 130 mm Hg and / or diastolic blood pressure (DBP) <60 mm Hg or ≥ 85 mm Hg;
14. Heart rate less than 60 beats/min or more than 90 beats/min at the time of screening, respiratory rate less than 12 or more than 18 per minute at the time of screening, body temperature below 36.0 ° C or above 37.0 ° C at the time of screening;
15. use of any prescription and ATC drugs:

    * including herbs and food additives, vitamins that can have a significant effect on the PK of rivaroxaban or data on the effect of which on the pharmacokinetics of rivaroxaban are unknown, as well as question the characterization of the volunteer as healthy, less than 14 days before taking the drug in the first period;
    * including the use of drugs that are inducers or inhibitors of isoenzymes CYP3A4, CYP2J2 (HIV protease inhibitors, antifungal drugs of the azole group, clarithromycin, erythromycin, phenytoin, carbamazepine, phenobarbital, St. John's wort preparations, etc.), less than 30 days before taking the drug in the first period;
16. donation of plasma or blood (450 ml or more) less than 2 months (60 days) before taking the drug in the first period;
17. consumption of caffeine and xanthine-containing drinks and products (tea, coffee, chocolate, cola, etc.), products containing poppy seeds, less than 48 hours before taking the drug in the first period;
18. consumption of alcohol and alcohol-containing foods and beverages less than 48 hours before taking the drug in the first period;
19. use of citrus fruits (including grapefruit and grapefruit juice) and cranberries (including juices, fruit drinks, etc.) less than 7 days before taking the drug in the first period;
20. intake of more than 10 units alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml dry wine or 50 ml of spirits) or history of alcoholism, drug addiction, drug abuse;
21. intense physical activity less than 24 hours before taking the drug in the first period;
22. smoking more than 10 cigarettes per day, including less than 24 hours before taking the drug in each period and during each study period;
23. participation in other clinical trials of drugs less than 3 months before taking the drug in the first period;
24. test positive for syphilis, hepatitis B, hepatitis C or HIV at the time of screening;
25. positive test for alcohol in exhaled air;
26. positive urinalysis for the content of narcotic and potent substances during screening (opiates, morphine, barbiturates, benzodiazepines, cannabinoids/marijuana);
27. the value of standard laboratory and instrumental parameters that go beyond the reference values;
28. lack of intention of volunteers to comply with the Protocol requirements throughout the course of the study and/or lack, in the opinion of the Investigator, of the volunteers' ability to understand and evaluate the information on this study as part of the informed consent form signing process, in particular regarding the expected risks and possible discomfort;
29. tattooing and piercing within 30 days prior to first drug administration;
30. difficulty swallowing tablets;
31. difficulty with taking blood (for example, difficult access to the veins).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-02-13 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Cmax of rivaroxaban in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00. 48.00 hours after each drug administration.
  Maximum observed concentration in plasma.
AUC0-t of rivaroxaban in plasma after administration of the test and the reference. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00. 48.00 hours after each drug administration.
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration using the linear trapezoidal method

SECONDARY OUTCOMES:
Tmax of rivaroxaban in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00. 48.00 hours after each drug administration.
  Time of maximum observed concentration; if it occurs at more than one time point, Tmax is defined as the first time point with this value.
AUC0-INF of rivaroxaban in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00. 48.00 hours after each drug administration.
  Area under the concentration time curve extrapolated to infinity, calculated as AUC0-t + ĈLQC (the predicted concentration at time TLQC) / λZ (apparent elimination rate constant).
Residual area of rivaroxaban in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00. 48.00 hours after each drug administration.
  Extrapolated area (AUCresid%=100%*(AUC0-INF - AUC0-t)/AUC0-INF).
λZ of rivaroxaban in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00. 48.00 hours after each drug administration.
  Apparent elimination rate constant.
Terminal elimination half-life (T1/2) of rivaroxaban in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00. 48.00 hours after each drug administration.
  Terminal elimination half-life, calculated as ln(2)/λZ.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Khokhlov, Principal Investigator — ClinPharmInvest, LLC
Locations (1):
- Private healthcare institution "Clinical Hospital "RZD-Medicine" of the city of Yaroslavl", Yaroslavl, Russia